CLINICAL TRIAL: NCT05791032
Title: Sub Chronic Evaluation for ATP With an Extravascular Placed ICD Lead (STEP ICD) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtaCor Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DOC-10246
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Ventricular Arrythmia; Ventricular Tachycardia; Ventricular Fibrillation
Keywords: Ventricular Defibrillation; Extravascular
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AtaCor EV-ICD Lead System (Experimental): Subjects implanted with the AtaCor EV-ICD Lead
  Interventions: Device: AtaCor EV-ICD Lead

INTERVENTIONS:
Device: AtaCor EV-ICD Lead — Subjects will receive the AtaCor EV-ICD Lead being evaluated in the study.

SUMMARY:
STEP ICD is a premarket, exploratory, early feasibility, interventional study designed to evaluate the preliminary safety and performance of the Investigational Devices. The study is intended to inform the final device design which will be further evaluated in traditional feasibility and /or pivotal clinical investigations.

The primary safety objective is to characterize safety of the EV-ICD Lead through 3 months post-implant. The primary performance objective is to characterize sensing and conversion of induced VF with the EV-ICD Lead up to 3 months post-implant.

DETAILED DESCRIPTION:
The primary safety endpoint is incidence of Adverse Device Effects (ADEs). The primary performance endpoint is induced VF conversion success up to 3 months post-implant. Secondary endpoints include defibrillation metrics (i.e., lowest Conversion Energy (J), ability to automatically sense and detect ventricular arrhythmias, detection time and time-to-therapy) and pacing metrics (ventricular capture threshold (V), pacing impedance (ohms), R-wave amplitude (mV), and extracardiac pacing sensation level).

Up to 30 eligible Subjects undergoing a pectoral transvenous ICD procedure (de novo or replacement) will receive an EV-ICD Lead connected to a commercially available ICD in a left mid-axillary or left pectoral pocket.

The EV-ICD System will be tested in the intended implant location to determine the lowest defibrillation energy. Subjects will remain in the hospital overnight (at a minimum), prior to discharge. Except during testing, the EV-ICD System will remain programmed to monitor only (therapy OFF) to detect and store ventricular arrhythmias over the follow-up period. A concomitantly implanted transvenous ICD (TV-ICD) system will provide any necessary ICD therapy. Non-therapy EV-ICD programming parameters will match the TV-ICD to the extent possible to facilitate recording of matched stored electrograms.

Follow-up visits are planned at pre-discharge, 2 weeks, 1 month, 2 months, and 3 months. VF conversion testing will occur prior to lead removal in order to test subchronic defibrillation effectiveness with a submaximal energy shock in standard and/or reverse polarity. At the Lead Removal Follow Up, the EV-ICD System will be explanted and the TV-ICD System left in place.

A final follow-up will occur one month after EV-ICD Lead explant to assess any post-explant adverse events prior to study exit.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Indicated for de novo or replacement ICD procedure

Exclusion Criteria:

1. BMI ≥ 35 kg/m2
2. Subjects who require continual ventricular pacing
3. Presence or planned use of a subcutaneous ICD lead, subcutaneous coils/arrays, epicardial patches or epicardial pace/sense leads within the study period
4. Planned MRI within the study period
5. Subjects on anticoagulation or antiplatelet therapy that cannot be temporarily discontinued for the procedure
6. Circumstances that may prevent data collection or follow-up
7. Participation in any concurrent clinical study without prior written approval from the Sponsor
8. Inability or unwillingness to provide informed consent to participate in the Study

   Known prior history for any of the following:
9. NYHA IV functional class in past 90 days
10. Inotropic therapy in past 180 days
11. Structural abnormalities of the heart that may increase risk of the study procedure or an obstructed/restricted pathway into the mediastinum
12. Uncontrolled paroxysmal, persistent or permanent atrial fibrillation
13. Median or partial sternotomy
14. Surgery with disruption of the lung, pericardium or connective tissue between the sternum and pericardium
15. Significant anatomic derangement of or within the thorax (e.g., pectus excavatum, significant scoliosis)
16. Thoracic radiation therapy, pneumothorax, pneumomediastinum or other medical treatments which may complicate the AtaCor EV-ICD Lead System implant procedure
17. Any conditions which may complicate the AtaCor EV-ICD Lead System implant procedure
18. Pericardial disease, pericarditis and mediastinitis
19. Medical treatments, surgeries or conditions that increase the potential for adhesions in the thorax
20. FEV1 < 1.0 Liter
21. Surgically corrected congenital heart disease (not including catheter-based procedures)
22. Allergies to the device materials as listed in the Instructions for Use (IFU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Incidence of ADEs | Up to 3 months post-implant
  Incidence of Adverse Device Effects (ADEs)
Induced VF Conversion Success | Up to 3 months post-implant
  Induced VF conversion success up to 3 months post-implant

CONTACTS AND LOCATIONS:
Overall Officials: Martin C Burke, DO, Principal Investigator — AtaCor Medical, Inc.
Locations (1):
- Sanatorio Italiano, Asunción, Paraguay

REFERENCES:
- [Derived] Doshi SK, Knops RE, Ebner A, Husby M, Marcovecchio A, Sanghera R, Scheck D, Burke MC. Evaluation of a second-generation intercostal extravascular implantable cardioverter defibrillator lead with a pectoral pulse generator for sensing, defibrillation, and anti-tachycardia pacing. Europace. 2025 Mar 5;27(3):euaf044. doi: 10.1093/europace/euaf044. PMID 40037337